CLINICAL TRIAL: NCT02958735
Title: Human Performance: Role of Acute Exercise in Enhancing Cognitive Function
Brief Title: Exercise and Cognition Trials
Acronym: EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00076336
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Alteration of Cognitive Function
Keywords: exercise; cognition; brain-derived neurotrophic factor; insulin-like growth factor 1; cortisol
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rest (No Intervention): Participants randomly assigned to this arm rest quietly for thirty minutes instead of participating in the exercise challenge.
- Mild Exercise (Experimental): Participants randomly assigned to this arm are made to maintain a heart rate equivalent to 60% of the heart rate observed when VO2 max was achieved in the maximal stress test from the first visit.
  Interventions: Other: Exercise Challenge
- Hard Exercise (Experimental): Participants randomly assigned to this arm are made to maintain a heart rate equivalent to 80% of the heart rate observed when VO2 max was achieved in the maximal stress test from the first visit.
  Interventions: Other: Exercise Challenge

INTERVENTIONS:
Other: Exercise Challenge — Participants randomized to an exercise condition will perform treadmill exercise for 30 minutes. Participants will self-select a comfortable walking speed. The treadmill grade will be adjusted to elicit and maintain the target heart rate.
  Arms: Hard Exercise; Mild Exercise

SUMMARY:
The purpose of this study is to determine whether an acute bout of exercise may temporarily enhance cognitive function (such as memory or attention span) by measuring behavioral performance on cognitive tests, as well as expression of hormones in circulation associated with brain plasticity and stress.

DETAILED DESCRIPTION:
This is a randomized experiment consisting of three visits for each participant. Participants are determined to be eligible beforehand during a phone screening, in which the various study inclusions and exclusions are determined and the Physical Activity Readiness Questionnaire for Everyone 2015 (PARQ) is administered.

In the first visit, various anthropometric data are collected from participants, such as height, weight, and waist and hip circumference. The participants' blood pressure is also checked for hypertension. The participants are given Dual Energy X-Ray Absorptiometry (DEXA) scans to determine total body composition (bone, fat, and fat-free mass) If the participant is female, a urine analysis to determine pregnancy is required during the visit before the DEXA to ensure safety. Participants are given the Rapid Assessment of Physical Activity (RAPA) questionnaire to assess habitual activity levels. The participants' muscle strength is also measured using the Biodex System 3, an isokinetic dynamometer. The participants then undergo a maximal stress test on a treadmill integrated with a Cardinal Health Metabolic/ECG cart using a modified Balke protocol, beginning at 3 mph, 0% grade, and increasing 2.5% grade every 3 minutes. The ECG component of the metabolic cart will be used for continuous heart rate monitoring as part of the fitness assessment. Cardiorespiratory parameters (VO2, ventilation, respiratory rate) will also be measured throughout the test. Blood pressure is measured during the last 30 seconds of each exercise stage and the rating of perceived exertion (RPE) using the Borg 6 to 20 scale is obtained during each stage. Subjects are urged to give a maximal effort and are pushed until volitional fatigue.

In the second visit, participants are first given a series of cognitive tests designed to quantify such cognitive faculties as visual short-term memory, selective attention, processing speed, and verbal fluency. These tests consist of seeing simple images on a computer screen, such as a series of colored shapes, and responding using a keypad. A blood sample is also collected from the participants to serve as a baseline. The subject is then randomized to one of three groups: the first group rests for 30 minutes; the second group walks on the treadmill at a mild intensity, defined as maintaining 60% of the heart rate observed during the max VO2 from the first visit; the last group walks on the treadmill at a hard intensity, defined as maintaining 80% of the heart rate observed during the max VO2 from the first visit. The subjects then undergo a second blood draw after cooling down, followed immediately by another round of the same cognitive tests. An hour after finishing the exercise intervention, the same procedure of blood draw followed by cognitive tests is repeated, and an hour after that it is repeated again.

The third visit must be about 24 hours after the previous visit. Participants have blood drawn and one final round of cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of between 18.5 and 35 kg/m2
* Normal or corrected-to-normal vision
* No contraindications to participation in moderate to hard intensity physical activity

Exclusion Criteria:

* Self-report of alcohol or substance abuse in the past year or current treatment
* Women who are pregnant or nursing
* BMI of < 18.5 or > 35 kg/m2
* Diabetes mellitus. Subjects will be excluded for diabetes even if controlled by medications
* Cigarette smoking in the previous 12 weeks
* Elevated blood pressure (BP) defined as systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg
* Self-report of cardiovascular disease, cancer, renal disease, and other serious conditions that could be exacerbated by moderate intensity physical activity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
visual short-term memory questionnaire | baseline
  participants are shown sets of colored squares briefly and must pick out the square that changed color after a delay, scored on accuracy (0-100%)
visual short-term memory questionnaire | up to 5 minutes post intervention
  participants are shown sets of colored squares briefly and must pick out the square that changed color after a delay, scored on accuracy (0-100%)
visual short-term memory questionnaire | 1 hour after intervention
  participants are shown sets of colored squares briefly and must pick out the square that changed color after a delay, scored on accuracy (0-100%)
visual short-term memory questionnaire | 2 hours after intervention
  participants are shown sets of colored squares briefly and must pick out the square that changed color after a delay, scored on accuracy (0-100%)
visual short-term memory questionnaire | 24 hours after baseline
  participants are shown sets of colored squares briefly and must pick out the square that changed color after a delay, scored on accuracy (0-100%)
visual long-term memory questionnaire | 24 hours after baseline
  participants encode images in a cover task at baseline, scored on accuracy (0-100%)
verbal fluency | baseline
  participants are asked to name as many words as they can that begin with a certain letter within 1 minute, scored on number of appropriate words
verbal fluency | up to 5 minutes post intervention
  participants are asked to name as many words as they can that begin with a certain letter within 1 minute, scored on number of appropriate words
verbal fluency | 1 hour after intervention
  participants are asked to name as many words as they can that begin with a certain letter within 1 minute, scored on number of appropriate words
verbal fluency | 2 hours after intervention
  participants are asked to name as many words as they can that begin with a certain letter within 1 minute, scored on number of appropriate words
verbal fluency | 24 hours after baseline
  participants are asked to name as many words as they can that begin with a certain letter within 1 minute, scored on number of appropriate words
cortisol in circulation | baseline
  in nanograms per milliliter (ng/ml)
cortisol in circulation | up to 5 minutes post intervention
  in nanograms per milliliter (ng/ml)
cortisol in circulation | 1 hour after intervention
  in nanograms per milliliter (ng/ml)
cortisol in circulation | 2 hours after intervention
  in nanograms per milliliter (ng/ml)
cortisol in circulation | 24 hours after baseline
  in nanograms per milliliter (ng/ml)
igf-1 in circulation | baseline
  insulin-like growth factor 1 in nanograms per milliliter (ng/ml)
igf-1 in circulation | up to 5 minutes post intervention
  insulin-like growth factor 1 in nanograms per milliliter (ng/ml)
igf-1 in circulation | 1 hour after intervention
  insulin-like growth factor 1 in nanograms per milliliter (ng/ml)
igf-1 in circulation | 2 hours after intervention
  insulin-like growth factor 1 in nanograms per milliliter (ng/ml)
igf-1 in circulation | 24 hours after baseline
  insulin-like growth factor 1 in nanograms per milliliter (ng/ml)
bdnf in circulation | baseline
  brain-derived neurotrophic factor in nanograms per milliliter (ng/ml)
bdnf in circulation | up to 5 minutes post intervention
  brain-derived neurotrophic factor in nanograms per milliliter (ng/ml)
bdnf in circulation | 1 hour after intervention
  brain derived neurotrophic factor in nanograms per milliliter (ng/ml)
bdnf in circulation | 2 hours after intervention
  brain-derived neurotrophic factor in nanograms per milliliter (ng/ml)
bdnf in circulation | 24 hours after baseline
  brain-derived neurotrophic factor in nanograms per milliliter (ng/ml)
general executive functioning as assessed by the stroop test questionnaire | baseline
  participants must identify the color of various words on the screen irrespective of their meaning, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the stroop test questionnaire | up to 5 minutes post intervention
  participants must identify the color of various words on the screen irrespective of their meaning, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the stroop test questionnaire | 1 hour after intervention
  participants must identify the color of various words on the screen irrespective of their meaning, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the stroop test questionnaire | 2 hours after intervention
  participants must identify the color of various words on the screen irrespective of their meaning, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the stroop test questionnaire | 24 hours after baseline
  participants must identify the color of various words on the screen irrespective of their meaning, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the flanker task questionnaire | baseline
  participants must identify the orientation of a central arrow while ignoring those of other arrows on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the flanker task questionnaire | up to 5 minutes post intervention
  participants must identify the orientation of a central arrow while ignoring those of other arrows on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the flanker task questionnaire | 1 hour after intervention
  participants must identify the orientation of a central arrow while ignoring those of other arrows on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the flanker task questionnaire | 2 hours after intervention
  participants must identify the orientation of a central arrow while ignoring those of other arrows on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the flanker task questionnaire | 24 hours after baseline
  participants must identify the orientation of a central arrow while ignoring those of other arrows on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the irrelevant capture task questionnaire | baseline
  participants must identify a set of symbols as either letters or numbers while ignoring distracting images that flash on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the irrelevant capture task questionnaire | up to 5 minutes post intervention
  participants must identify a set of symbols as either letters or numbers while ignoring distracting images that flash on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the irrelevant capture task questionnaire | 1 hour after intervention
  participants must identify a set of symbols as either letters or numbers while ignoring distracting images that flash on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the irrelevant capture task questionnaire | 2 hours after intervention
  participants must identify a set of symbols as either letters or numbers while ignoring distracting images that flash on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds
general executive functioning as assessed by the irrelevant capture task questionnaire | 24 hours after baseline
  participants must identify a set of symbols as either letters or numbers while ignoring distracting images that flash on the screen, scored based on accuracy (0-100%) and reaction time in milliseconds

SECONDARY OUTCOMES:
total and regional bone mass | baseline
  as assessed by dual-energy x-ray absorptiometry (DEXA) scan, in grams per square centimeter (g/cm2)
total and regional fat and fat-free mass | baseline
  as assessed by dual-energy x-ray absorptiometry (DEXA) scan in grams per square centimeter (g/cm2)
habitual activity levels | baseline
  as assessed by Rapid Assessment of Physical Activity questionnaire, possible scores are: Active, Under Active Regular, Under Active Regular- Light Activities, Under Active, Sedentary
muscle strength | baseline
  as measured by isokinetic testing using the Biodex System 3
cardiorespiratory endurance | baseline
  as assessed by maximal stress test, represented by heart rate at maximal oxygen uptake
body mass index (BMI) | baseline
  measured in kilograms per square meter (kg/m2)
waist-to-hip ratio | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stewart, EdD, Principal Investigator — Johns Hopkins University; Peter Searson, PhD, Principal Investigator — Johns Hopkins University; Howard Egeth, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No